CLINICAL TRIAL: NCT02265367
Title: Novel Medication as a Potential Smoking Cessation Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 1409M53561
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Results first posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-03

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Levomilnacipran

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levomilnacipran (Experimental): In the first three week period levomilnacipran is evaluated whereas in the second three week period placebo is evaluated
  Interventions: Drug: Levomilnacipran; Drug: Placebo
- Placebo (Experimental): In the first three week period placebo is evaluated whereas in the second three week period levomilnacipran is evaluated
  Interventions: Drug: Levomilnacipran; Drug: Placebo

INTERVENTIONS:
Drug: Levomilnacipran
  Other Names: Fetzima
Drug: Placebo

SUMMARY:
The purpose of this study is to provide preliminary information assessing if levomilnacipran may be effective at increasing smoking cessation rates.

ELIGIBILITY:
Inclusion Criteria:

* Be between 25 years old and 55 years old
* Smoke a minimum number of cigarettes per day
* Indicate motivation to quit smoking

Exclusion Criteria:

* Current or history of medical or psychiatric conditions that could interfere with measures being studied or that could be affected by the study medication
* Use of medication that could interfere with measures to be studied or that could be expected to interact with levomilnacipran
* Are pregnant or breast feeding

The investigators will evaluate if there are other reasons why someone may not be eligible to participate

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2015-01; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kotlyar, PharmD, Principal Investigator — University of Minnesota
Locations (1):
- Clinical and Translational Sciences Institute, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Levomilnacipran Then Placebo: In the first three week period, baseline measures are obtained during the first week, levomilnacipran started during the second week and effects on smoking behavior assessed during the third week. For the subsequent three-week period, washout occurs during the first week, placebo is started during the second week and effects on smoking behavior assessed during the third week.
- Placebo Then Levomilnacipran: In the first three week period, baseline measures are obtained during the first week, placebo started during the second week and effects on smoking behavior assessed during the third week. For the subsequent three-week period, washout occurs during the first week, levomilnacipran is started during the second week and effects on smoking behavior assessed during the third week.
  Placebo
Period: Overall Study
Arm/Group | Levomilnacipran Then Placebo | Placebo Then Levomilnacipran
Started | 28 | 28
Completed First 3-week Period | 24 | 26
Completed (Completer defined as participants who completed at least 2 of the 5 assessments occurring during the third week of each three-week period.) | 18 | 22
Not Completed | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- Placebo Then Levomilnacipran: In the first three week period, baseline measures are obtained during the first week, placebo started during the second week and effects on smoking behavior assessed during the third week. For the subsequent three-week period, washout occurs during the first week, levomilnacipran is started during the second week and effects on smoking behavior assessed during the third week.
- Total: Total of all reporting groups
Arm/Group | Levomilnacipran Then Placebo | Placebo Then Levomilnacipran | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Full Range); unit: Years] | 45 [28 to 55] | 44 [26 to 55] | 44 [26 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 19 | 21 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 25 | 26 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 8 | 20
  White | 14 | 16 | 30
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Percent of Days of Confirmed Abstinence (Out of 5 Maximum)
Description: Subjects will be asked to abstain for five consecutive days during the third week of each intervention period with the percentage of confirmed abstinence days being the primary outcome measure
Time Frame: 5 days
Population: Only participants who completed the study were analyzed. Completers were those with data from at least 2 days during the third week of the second three week period
Measure: Mean (Standard Error); unit: percentage of days non-smoking
Groups:
- Levomilnacipran: In this three week period, baseline measures are obtained during the first week, levomilnacipran started during the second week and effects on smoking behavior assessed during the third week.
- Placebo: In this three week period, baseline measures are obtained during the first week, placebo during the second week and effects on smoking behavior during the third week
Arm/Group | Levomilnacipran | Placebo
Number analyzed (Participants) | 40 | 40
percentage of days non-smoking | 46.9 (6.7) | 42.0 (6.5)

ADVERSE EVENTS:
Time Frame: Adverse events that were reported during the period (up to 2 weeks) when participants were taking either levomilnacipran or placebo
Description: Participants were asked to report any side effects or health changes that occurred regardless of whether they thought that these were related to the study medication
Groups:
- Levomilnacipran: In this three week period, baseline measures are obtained during the first week, levomilnacipran will be started during the second week and effects on smoking behavior will be assessed during the third week
  Levomilnacipran
- Placebo: In this three week period, baseline measures are obtained during the first week, placebo will be started during the second week and effects on smoking behavior will be assessed during the third week
  Placebo
Arm/Group | Levomilnacipran | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 37/52 | 26/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levomilnacipran (N=52) | Placebo (N=51)
Sleep / Energy Changes (General disorders) | 16 | 12
Gastrointestinal Symptoms (Gastrointestinal disorders) | 11 | 10
Headache (General disorders) | 9 | 8
Changes in Mood, Anxiety or Irritability Level (Psychiatric disorders) | 7 | 2
Dizziness (General disorders) | 1 | 5
Excessive Sweating (General disorders) | 3 | 3
Body aches / pains (Musculoskeletal and connective tissue disorders) | 4 | 2
Dry mouth (General disorders) | 3 | 2
Change in Appetite (Gastrointestinal disorders) | 3 | 2
Cold / Seasonal Allergy Symptoms (Respiratory, thoracic and mediastinal disorders) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT02265367/Prot_SAP_000.pdf